CLINICAL TRIAL: NCT02595788
Title: Haemodynamic Changes During Anaesthesia in the Prone Position, Evaluated Using Transoesophageal Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Joachim Torp Hoffmann-Petersen, MD, Odense University Hospital
Other Study IDs: S-20130032
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Spinal Surgery; Anaesthesia; Changes in Left and Right Ventricle Dimension; Changes in Bloodflow Across Cardiac Valves; Changes in Dimensions of Inferior Caval Dimension and Hepatic Venous Bloodflow; Changes i Myocardial Velocities; Changes in Diastolic Function
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Supine position: Examination in the supine position
- Prone position: Change from supine to prone position
  Interventions: Other: Change from supine to prone position

INTERVENTIONS:
Other: Change from supine to prone position — Change from supine to prone position
  Groups: Prone position

SUMMARY:
Transoesophageal ultrasound examination before and after prone position.

DETAILED DESCRIPTION:
Patients undergoing spinal surgery in the prone position are anaesthetized and then an ultrasound probe is placed in the oesophagus and the heart physiology is examined. Following prone position the examination is repeated.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for spinal surgery in the prone position. Body mass index above 30.

Exclusion Criteria:

* significant cardiomyopathy or valvular disease
* heart rhythm other than normal sinus rhythm
* coagulopathy
* increased risk of oesophageal injury during probe insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for spinal surgery in the prone position. Body mass index above 30.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
End systolic and diastolic dimension of the left and right ventricle. | The day of surgery
  Studied after induction of anaesthesia, before and after the patient is placed in the prone position.

SECONDARY OUTCOMES:
Left and rigth ventricle eccentricity index. | The day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Hoffmann-Petersen, MD, Principal Investigator — Specialist Registrar
Locations (1):
- Odense University Hospital, Odense, Denmark